CLINICAL TRIAL: NCT06230679
Title: Effectiveness of NESA in the Treatment of Sleep Problems, Fatigue, and Neuromuscular Pain in Cancer Survivors.
Brief Title: Effectiveness of NESA in the Treatment of Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aníbal Báez Suárez (Other)
Responsible Party: Sponsor-Investigator, Aníbal Báez Suárez, Clinical Professor, University of Las Palmas de Gran Canaria
Organization: University of Las Palmas de Gran Canaria (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NESABiel
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-08

CONDITIONS: Cancer Survivors
Keywords: cancer; physical therapy modality; Electric Stimulation Therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive Neuromodulation (Experimental): Intervention with electrical stimulation: application of 6 electrodes per extremity and an adhesive electrode at C7 level.
  Interventions: Device: Non-invasive Neuromodulation
- Placebo Non-invasive Neuromodulation (Placebo Comparator): Intervention with electrical stimulation: application of 6 electrodes per extremity and an adhesive electrode at C7 level.
  Interventions: Device: Placebo Non-invasive Neuromodulation

INTERVENTIONS:
Device: Non-invasive Neuromodulation — Patients receive non-invasive neurostimulation through the Nesa device
  Arms: Non-invasive Neuromodulation
Device: Placebo Non-invasive Neuromodulation — The same protocol described for the experimental group will be applied, but electrical stimulation device which will be previously manipulated and tested with an oscilloscope so that they do not emit electrical currents.
  Arms: Placebo Non-invasive Neuromodulation

SUMMARY:
Cancer is a disease, or a set of diseases, that increased in our society. However, improvements in their detection and treatment increase the number of patients who survive. Every year 2.6 million people are diagnosed in the European Union and 1.4 million become cancer survivors. However, these people suffer the late adverse effects of treatment that can seriously affect their quality of life.

the most common late effects are pain, fatigue, and sleeping difficulties. These are estimated between 58-90%. The autonomic nervous system (ANS) appears to play an important role in the manifestation and perpetuation of these symptoms.

DETAILED DESCRIPTION:
This study aims to evaluate NESA (or NESA non-invasive neuromodulation) to treat the most common long-term side effects in cancer survivors, due to the most used treatments.

It will be compared between two groups of cancer survivors. The intervention group, with electrical stimulation, and the sham group, without electrical stimulation emission. The subjects will be assigned randomly. Neither the patient, the therapist, nor the analysts/researchers will know the assignment.

Finally, this project aims to add a passive tool to the therapeutic arsenal of health professionals in the oncology field for the treatment of late side effects.

ELIGIBILITY:
Inclusion Criteria:

* Be a cancer survivor (5 years after discharge)
* Have 1 of the 3 symptoms of the most common cluster: sleep problems, chronic fatigue, chronic neuro-muscular pain.

Exclusion Criteria:

* Not have an active oncological process
* Present any of the contraindications of the NESA-XSignal device: pacemaker, internal bleeding, skin in poor condition (ulcerations or wounds), acute febrile processes, acute thrombophlebitis, pregnancy, phobia of electricity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality assessed by Pittsburgh Sleep Quality Index (PSQI) | Measurement of change: before treatment (baseline), at two months (end of treatment), and at 1 months of treatment (follow-up period).
  The investigators want to see if there are improvements in the quality, efficiency, and quantity of sleep. The Pittsburgh Sleep Quality Index (PSQI) will be combined to report changes in the patient's sleep quality.
  Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
  Adding up the average scores of the seven factors gives a global PSQI score from 0 to 21, with 0-4 indicating "good" sleep and 5-21 indicating "poor" sleep
Change in quality of life assessed by The Short Form 36 (SF-36) health questionnaire | Measurement of change: before treatment (baseline), at two months (end of treatment), and at 1 months of treatment (follow-up period).
  The Short Form 36 (SF-36) health questionnaire will be used. It is a generic scale that provides a profile of health status and is applicable to both patients and the general population.
  It is composed of 36 questions (items) that assess both positive and negative states of health. The scores for each of the 8 dimensions of the SF-36 range from 0 to 100, with 100 indicating optimal health and 0 reflecting very poor health.
Change in Pain assessed by McGill Pain questionnaire | Measurement of change: before treatment (baseline), at two months (end of treatment), and at 1 months of treatment (follow-up period).
  It is a self-report questionnaire that allows to give a good description of the quality and intensity of the pain they are experiencing. of the quality and intensity of the pain they are experiencing. It consists of a list of 78 words in 20 sections related to pain. Users mark the words that best describe their pain. users mark the words that best describe their pain. These words correlate with different aspects of pain different aspects of pain, including a sensory section (sections 1 to 10), an affective section (sections 11 to 15), an evaluative section (sections 11 to 15), and a 10), an affective section (sections 11 to 15), an evaluative section (section 16), and finally a miscellaneous section (section 16). and, finally, a miscellaneous section (sections 17 to 20).
  The main component of the McGill Pain questionnaire consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Amengual Jaume, MSc, Principal Investigator — University of Las Palmas de Gran Canaria
Locations (1):
- Gutmotion, Santa Maria del Camí, Balearic, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rick O, Dauelsberg T, Kalusche-Bontemps EM. Oncological Rehabilitation. Oncol Res Treat. 2017;40(12):772-777. doi: 10.1159/000481709. Epub 2017 Nov 29. PMID 29183040
- [Result] Paltrinieri S, Fugazzaro S, Bertozzi L, Bassi MC, Pellegrini M, Vicentini M, Mazzini E, Costi S. Return to work in European Cancer survivors: a systematic review. Support Care Cancer. 2018 Sep;26(9):2983-2994. doi: 10.1007/s00520-018-4270-6. Epub 2018 May 29. PMID 29845421
- [Result] Boland EG, Ahmedzai SH. Persistent pain in cancer survivors. Curr Opin Support Palliat Care. 2017 Sep;11(3):181-190. doi: 10.1097/SPC.0000000000000292. PMID 28700361
- [Result] Kline-Quiroz C, Nori P, Stubblefield MD. Cancer Rehabilitation: Acute and Chronic Issues, Nerve Injury, Radiation Sequelae, Surgical and Chemo-Related, Part 1. Med Clin North Am. 2020 Mar;104(2):239-250. doi: 10.1016/j.mcna.2019.10.004. Epub 2019 Nov 23. PMID 32035566